CLINICAL TRIAL: NCT05324696
Title: Autoinflation: Alternative in the Treatment of Otitis Media With Effusion
Acronym: OME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Ciências Biomédicas Abel Salazar (Other)
Responsible Party: Principal Investigator, Joao Lino, Principal Investigator, Instituto de Ciências Biomédicas Abel Salazar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 052-DEFI/ 053-CE
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-04

CONDITIONS: Otitis Media With Effusion; Hearing Loss
MeSH Terms: conditions — Otitis Media with Effusion; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment with placebo device (Placebo Comparator): Device similar to the one developed, but which does not generate pressure
  Interventions: Device: autoinflation device
- Treatment with a working device (Experimental): Treatment with a functioning device, which generates the necessary pressure to open the Eustachian tube
  Interventions: Device: autoinflation device
- Surgical treatment (Active Comparator): Surgical treatment (myringotomy with placement of ventilation tubes) which is the treatment currently applied in children with otitis media with effusion that do not resolve with medical treatment and/or autoinflation
  Interventions: Device: autoinflation device

INTERVENTIONS:
Device: autoinflation device — The authors developed a new standardized, inexpensive and simple device, based on Moniri. The Device is formed by a T tube with a unidirectional valve. A mask with the capacity of covering the child's mouth and nose, providing hermetic seal, and a balloon are connected to 2 ends of the T tube. Blowing the balloon trough the mask, with different types of maneuvers, will force the opening of the Eustachian tube and subsequent reabsorption of the middle ear effusion.

SUMMARY:
Otitis media with effusion (OME) is a common finding affecting children and the main cause of acquired hearing loss in the pediatric age.

OBJECTIVES

The purpose of the clinical study is to determine whether self-inflation using a new device:

* It is an effective non-invasive treatment during the watchful waiting period, with the ability to improve hearing loss and prevent surgical treatment;
* Maintains long-term hearing improvement;

DETAILED DESCRIPTION:
1. Introduction

   Otitis media with effusion (OME) is a common finding affecting children in the age of 2-6 years. Although OME is the main cause of acquired hearing loss in the pediatric age, it's treatment it's still controversial. Due to high spontaneous resolution, current international guidelines recommend a period of "watchful waiting" for 3 to 6 months after which, if the hearing loss persists, surgery with tympanostomy tube insertion under general anesthesia is indicated.

   During the watchful waiting period, medical treatment options, such as oral and nasal corticosteroids, antibiotics, mucolytics or nasal decongestants, are not recommended due to lack of effect or side effects. Nevertheless, the results of autoinflation in the treatment of OME in children are divergent although suggestive of clinical effect in the short-term.

   In a previous study the authors concluded that autoinflation with a new device - Moniri® Medical Device - resolved the OME and prevented surgery in 80% of children with chronic OME.

   In this study, the authors developed a new standardized, inexpensive and simple device, based on Moniri® Medical Device. The Device is formed by a T tube with a unidirectional valve. A mask with the capacity of covering the child's mouth and nose, providing hermetic seal, and a balloon are connected to 2 ends of the T tube. Blowing the balloon trough the mask, with different types of maneuvers, will force the opening of the Eustachian tube and subsequent reabsorption of the middle ear effusion.
2. Aime Our aim it's to prove that autoinflation is an efficient non-invasive treatment during the watchful waiting period, with the capacity of improving hearing loss thus preventing surgical treatment.
3. Material and Methods

   * Study design:

   Clinical investigation, prospective, blinded and randomized.
   * Sample:

   Children between 3 and 8 years of age

   - Inclusion criteria: Children between 3 and 8 years of age with otomicroscopic alterations suggestive of unilateral or bilateral OME; type B or C2 tympanogram (pressure ≤ 200 daPa); audiogram with hearing loss ≥ 20 dB or air-bone gap at the time of evaluation by an otolaryngologist.

   - Exclusion criteria: Children with uncontrolled asthma, craniofacial anomalies, active ear disease (retraction pouch, adhesive otitis or tympanic perforation) or a history of ear surgery.

   - Recruitment: Children followed up at the Otorhinolaryngology outpatient clinic at Centro Hospitalar do Porto with a diagnosis of OME, who are in watchful waiting period. Parents/legal guardians of children who meet the inclusion criteria are invited to participate.

   - Study groups

   Blindly and randomly, three study groups are created:

   > GROUP A: Treatment with placebo device

   > GROUP B: Treatment with a functioning device

   The Device to be studied results from the combination of different components, all of them used in different medical areas and all of them individually already approved by the National Authority for Medicines and Health Products. After an exposure to two expertises of the National Authority for Medicines and Health Products in the field of medical devices, the researchers were informed that the use of the combination of the various components should be considered an off-label use of the same and, as such, does not require formal requirement for approval of use.

   > GROUP C: Surgical treatment. Children undergoing surgical treatment for OME (myringotomy with placement of transtympanic ventilation tubes +/- adenoidectomy), as they have already exceeded the period of "watchful waiting" and who had a surgical indication, will be included in group C. This group, representative of the current treatment recommended in cases of persistent OME, will serve to compare results with the proposed new treatment.

   Study groups will be evaluated at 1, 3, 6, 12 and 18 months after treatment initiation (placebo device, functioning device or surgery).

   Children will undergo audiological assessment with otomicroscopy, tympanogram and audiogram. The results will be compared in the same child, to evaluate if there was resolution of OME, and between groups to evaluate the effectiveness of the treatments.

ELIGIBILITY:
- Inclusion criteria: Children between 3 and 8 years of age with otomicroscopic alterations suggestive of unilateral or bilateral OME; type B or C2 tympanogram (pressure ≤ 200 daPa); audiogram with hearing loss ≥ 20 dB or air-bone gap at the time of evaluation by an otolaryngologist.

- Exclusion criteria: Children with uncontrolled asthma, craniofacial anomalies, active ear disease (retraction pouch, adhesive otitis or tympanic perforation) or a history of ear surgery.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
Otitis media with effusion resolution proven with normalization of results in the audiological study (tympanogram and audiogram) | 3 years
  Outcomes assessed by sustained improvement in the audiological study carried out with the following complementary diagnostic tests: audiogram and tympanogram

CONTACTS AND LOCATIONS:
Overall Officials: João Lino, MD, Study Director — Instituto de Ciências Biomédicas Abel Salazar
Locations (1):
- Centro Hospitalar Univrsitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No